CLINICAL TRIAL: NCT01040455
Title: Therapeutic Response to Lansoprazole Among Different Subgroups of Functional Dyspepsia: a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Lansoprazole for Subgroups of Functional Dyspepsia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: failure to recruit enough patients
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200907053M
Record Dates: First submitted 2009-12-25; First posted 2009-12-29 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Functional Dyspepsia
Keywords: functional dyspepsia; lansoprazole; placebo effect
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lansoprazole (Experimental): lansoprazole 15mg (Takepron®, Takeda Pharmaceutical Company, Osaka, Japan) once daily for eight weeks
  Interventions: Drug: Lansoprazole
- placebo (Placebo Comparator): placebo once daily for eight weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lansoprazole — lansoprazole 15mg (Takepron®, Takeda Pharmaceutical Company, Osaka, Japan) once daily for eight weeks
  Other Names: Takepron
  Arms: lansoprazole
Drug: placebo — placebo once daily for eight weeks
  Arms: placebo

SUMMARY:
Pharmacotherapy for functional dyspepsia remains unsatisfactory. Previous randomized trials reported conflicting results on clinical effectiveness of proton pump inhibitor in patients with functional dyspepsia. This study aims to examine whether lansoprazole 15mg is more effective than placebo for functional dyspepsia in Taiwanese patients, and to investigate the association between subgroups of patients and therapeutic response.

DETAILED DESCRIPTION:
This is a prospective double-blind randomized placebo-controlled trial. A total of 450 dyspeptic adult patients, who are diagnosed with functional dyspepsia in accordance with Rome III criteria, are randomly allocated in a 1:1 proportion to receive either lansoprazole 15mg or placebo once daily for 8 weeks. Primary outcome is complete relief of dyspeptic symptoms. Secondary outcomes include significant symptomatic relief, improvement of dyspepsia severity, and health-related quality of life. We use a multiple logistic regression analysis to investigate whether dyspepsia subgroups are associated with different therapeutic responses.

ELIGIBILITY:
Inclusion Criteria:

* Dyspeptic adult outpatients
* Characteristic dyspeptic symptoms according to Rome III criteria (bothersome postprandial fullness, early satiation, epigastric pain, or epigastric burning)
* Upper gastrointestinal endoscopy excluding structural diseases

Exclusion Criteria:

* aged less than 20 years old,
* organic lesions such as peptic ulcer, tumor of any kind, stricture or structural deformity, erosive esophagitis, or vasculopathy on endoscopy
* typical and predominant reflux symptoms (heartburn or acid regurgitation)
* comorbidity with malignancy, diabetes mellitus, liver cirrhosis, renal failure, or porphyria
* history of intra-abdominal surgery
* concurrent use of aspirin, non-steroidal anti-inflammatory drug or proton pump inhibitor
* history of allergy or severe side effects to lansoprazole
* pregnant or lactating women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
complete relief of dyspeptic symptoms | within one week after complete study medication

SECONDARY OUTCOMES:
satisfactory therapeutic response (complete or marked relief of symptoms) | within one week after complete study medication
change of dyspepsia severity as measured by total scores of Hong Kong index | within one week after completing study medication
health-related quality of life as reflected in every aspect of SF-36 | within one week after completing study medication

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, M.D.,Ph.D., Principal Investigator — National Taiwan University College of Medicine
Locations (4):
- Taiwan (4):
  - National Taiwan University Hospital Yun-Lin Branch, Douliu
  - E-Da Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Veterans General Hospital-Taipei, Taipei

REFERENCES:
- [Background] Hsu YC, Liou JM, Liao SC, Yang TH, Wu HT, Hsu WL, Lin HJ, Wang HP, Wu MS. Psychopathology and personality trait in subgroups of functional dyspepsia based on Rome III criteria. Am J Gastroenterol. 2009 Oct;104(10):2534-42. doi: 10.1038/ajg.2009.328. Epub 2009 Jun 16. PMID 19532128
- See also: Rome Foundation — http://www.romecriteria.org/